CLINICAL TRIAL: NCT06491459
Title: Predicting Postoperative Pulmonary Infection in Elderly Patients Undergoing Major Surgery: a Study Based on Logistic Regression and Machine Learning Models
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: UHCT21772
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pulmonary Infection in Elderly Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although a number of clinical predictive models were developed to predict postoperative pulmonary infection, few predictive models have been used in elderly patients. In this study, the researchers aim to compare different algorithms to predict postoperative pulmonary infection in elderly patients and to assess the risk of postoperative pulmonary infection in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 65 years
2. patients who were mechanically ventilated under major surgery

Exclusion Criteria:

1. preoperative tracheal intubation
2. preoperative pneumonia
3. organ transplantation
4. missing data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients underwent surgery at the tertiary hospital Hospital from January 2014 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 9481 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative pulmonary infection during hospitalization | through study completion, an average of 30 days
  the incidence of postoperative pulmonary infection during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Liu J, Li X, Wang Y, Xu Z, Lv Y, He Y, Chen L, Feng Y, Liu G, Bai Y, Xie W, Wu Q. Predicting postoperative pulmonary infection in elderly patients undergoing major surgery: a study based on logistic regression and machine learning models. BMC Pulm Med. 2025 Mar 19;25(1):128. doi: 10.1186/s12890-025-03582-4. PMID 40108569